CLINICAL TRIAL: NCT03625934
Title: Study to Evaluate the Induction of HBV Virus Neutralizing Antibodies in Healthy Vaccine Naive Adults and Non-responders and in Patients Chronically Infected With HBV Using VVX001
Brief Title: Study to Evaluate Induction of HBV Virus Neutralizing Antibodies Using VVX001
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Viravaxx AG (Industry)
Collaborators: Gouya Insights (Unknown); KKS MedUni Vienna (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVX001-CS001
Record Dates: First submitted 2018-07-02; First posted 2018-08-10 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VVX001 (20 micrograms) (Experimental): Subjects will receive 5 injections of 20 micrograms each over a period of 4 months
  Interventions: Biological: VVX001
- Placebo (Placebo Comparator): Subjects will receive 5 s.c. injections of matching placebo over a period of 4 months
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VVX001 — 5 s.c. injections of 20 micrograms of VVX001 four weeks apart
  Arms: VVX001 (20 micrograms)
Biological: Placebo — 5 s.c. injections of matching Placebo four weeks apart
  Arms: Placebo

SUMMARY:
The Study will evaluate the effects of VVX001, a novel vaccine for hepatitis B, to

* elicit a robust protective IgG immune response in vaccine naive subjects
* in subjects who failed to demonstrate seroconversion after treatment with a licensed hepatitis B vaccine and
* in patients chronically infected with HBV.

DETAILED DESCRIPTION:
VVX001 is a recombinant fusion Protein composed of PreS from the large surface antigen of HBV and Peptides derived from the grass pollen allergen Phl p 5. In a previous trial in allergic but otherwise healthy subjects the product has been shown to elicit a potent IgG response to the epitope of PreS1, which is responsible for binding to the cellular receptor NTCP. These antibodies prevent infection with HBV in a cell culture model. The present study will evaluate if such an immune response can also be achieved in four different patient populations: 1) vaccine naive subjects; 2) subjects having failed to seroconvert upon vaccination with a licensed HBV vaccine; 3) patients who are chronically infected with HBV, but are classified as inactive carriers; 4) patients with active chronic HBV infection who are HbEAg negative and chronically treated with nucleo(t)side (NUC) antiviral drugs. All subjects will receive 5 s.c. injections of VVX001, the time course of antibody response to PreS1 will be monitored in all of them. In cohort 4) NUC treatment will be withdrawn at different timepoints during the study and the effect of treatment with VVX001 on hepatitis B disease Parameters will be monitored. Subjects will be followed for 6 months after the of treatment for Evaluation of a long-term effect.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: hepatits B vaccine naive subjects Seronegative for anti-HBs and anti-HBc antibodies and for HBs Antigen
* Cohort 2: Subjects who failed to develop a protective immune response upon standard vaccination with a licensed hepatitis B vaccine (<10 IU/L anti HbS antibodies) Seronegative for anti-HbS (<10 IU/L) and anti-HBc antibodies and for HbSAg
* Cohort 3: Parameters confirmed at screening during the past 12 months

  1. HBeAg negative;
  2. HbSAg positive at screening <3000 IU/ml;
  3. HBV viral load <2000 IU/ml
  4. ALT Levels ≤ULN at screening
* Cohort 4a: Parameters confirmed at screening during the last 12 months

  1. HBeAg negative;
  2. HbSAg positive <1000 IU/ml
  3. HBV DNA not detectable for at least 2 years
  4. History of nucleos(t)die Treatment for at least 3 years
  5. Willingness to discontinue NUC treatment during study
  6. ALT levels ≤ULN at screening
* Cohort 4b: in addition to cohort 4a:

  1. willingness to discontinue NUC treatment 6 weeks before entering the Study
  2. ALT Levels ≤ULN 6 weeks before entering the study and

     * 5x ULN at screening

Exclusion Criteria:

* Pregnant or breast-feeding females, adequate contraception required during the treatment phase
* History of grass pollen allergy
* Co-infection with HCV, HDV, HIV
* History of auto-immune hepatitis
* Elevated Levels of Alpha-Fetoprotein (AFP) >100 ng/ml
* Documented history of decompensated liver disease (albumin <3.5 g/dl and bilirubin >1.3 mg/dl)
* Autoimmune disorders, transplant recipients, use of immunosuppressive or immune modulating agents
* Oral corticosteroids of 20 mg/week within the past 4 weeks prior to screening
* History of treatment with PEG-IFN of IFN for at least 1 year prior to screening
* History of evidence or conditions associated with chronic liver disease
* Acute fever at time of enrolment
* History of alcohol abuse
* Planned administration of a vaccine not foreseen by study protocol in the period starting 30 days before first product administration and during the entire study period with exception of influenza vaccine
* History of Cancer
* Other severe co-morbid conditions and concurrent medication making the subject unsuitable for participation
* blood or plasma donation within 1 month of study enrolement and during the course of the study
* For all patients with chronic HBV infection:

  1. Total bilirubin >2x ULN confirmed by repeat testing within 2 weeks, unless historical documentation of Gilbert's syndrome
  2. Documented or suspected hepatocelluar carcinoma
  3. Presence of cholangitis, cholecystitis or bile duct obstruction
  4. Liver cirrhosis assessed by fibroscan with elastography <9kPa within the previous 12 months and FIB-score <3.2 at study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
PreS specific IgG antibodies | 4 weeks after the last injection of study drug
  Titer of PreS specific IgG antibodies

SECONDARY OUTCOMES:
PreS specific IgG, IgG1 and IgG4 antibodies | 4 weeks and 6 months after the last injection of study drug
  Titers of PreS specific IgG, IgG1 and IgG4 antibodies
HbSAg specific antibodies | 4 weeks and 6 months after the last injection of study drug
  Titers of HbSAg specific antibodies
Suppression of HBV infection | 4 weeks and 6 months after the last injection of study drug
  Suppression of HBV infection in HepG2-NTCP cells using HBV strain D3 in cell culture with patient sera
T cell proliferation | 4 weeks and 6 months after the last injection of study drug
  Proliferation of PreS specific CD4 and CD8 T cells
HbSAg titers | 4 weeks and 6 months after the last injection of study drug
  HbS Antigen titers will be measured in chronically infected patients
HBV DNA load | 4 weeks and 6 months after the last injection of study drug
  HBV DNA load will be measured by PCR in chronically infected patients
HBVcrAg titers | 4 weeks and 6 months after the last injection of study drug
  HBVcrAG titers will be measured in chronically infected patients

OTHER OUTCOMES:
Adverse events | up to 52 weeks
  Frequency, intensity and relatedness of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Petra Munda, MD, Principal Investigator — Medical University Vienna
Locations (2):
- Austria (2):
  - Medical University of Graz, Graz
  - Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cornelius C, Schoneweis K, Georgi F, Weber M, Niederberger V, Zieglmayer P, Niespodziana K, Trauner M, Hofer H, Urban S, Valenta R. Immunotherapy With the PreS-based Grass Pollen Allergy Vaccine BM32 Induces Antibody Responses Protecting Against Hepatitis B Infection. EBioMedicine. 2016 Sep;11:58-67. doi: 10.1016/j.ebiom.2016.07.023. Epub 2016 Aug 8. PMID 27568223
- [Background] Tulaeva I, Cornelius C, Zieglmayer P, Zieglmayer R, Schmutz R, Lemell P, Weber M, Focke-Tejkl M, Karaulov A, Henning R, Valenta R. Quantification, epitope mapping and genotype cross-reactivity of hepatitis B preS-specific antibodies in subjects vaccinated with different dosage regimens of BM32. EBioMedicine. 2020 Sep;59:102953. doi: 10.1016/j.ebiom.2020.102953. Epub 2020 Aug 24. PMID 32855110
- See also: Sponsor website — http://www.viravaxx.com